CLINICAL TRIAL: NCT05445427
Title: Outcomes of Treatment With Vagal Nerve Stimulation in Post-COVID Syndrome: A Pilot Study
Brief Title: Vagal Nerve Stimulation for Post COVID Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ryan T. Hurt, M.D., Ph.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-000925
Record Dates: First submitted 2022-07-01; First posted 2022-07-06 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Post COVID Syndrome; Fatigue; Headache
MeSH Terms: conditions — Fatigue; Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- VNS Treatment (Experimental): Subjects with post COVID syndrome with fatigue and headache will have vagal nerve stimulator applied to the neck for 2 minute intervals with two sets administered three times daily
  Interventions: Device: vagal nerve stimulator
- Non-VNS Treatment (No Intervention): Subjects with post COVID syndrome with fatigue and headache will receive current standard of care

INTERVENTIONS:
Device: vagal nerve stimulator — Non-invasive vagus nerve stimulator
  Arms: VNS Treatment

SUMMARY:
The purpose of this study is to evaluate the impact of vagal nerve stimulation on patients with post COVID syndrome who have fatigue and headache.

DETAILED DESCRIPTION:
Patients, after consenting, will perform questionnaires, have a blood samples taken, and undergo PET/CT scans of the brain. Patients will then be randomized to either receive vagal nerve stimulation, or continue standard clinical care. For those randomized to receive treatment, they will be given a device and asked to follow a specific regimen daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Presence of fatigue and post exertional malaise.
* Presence of headache
* Clinical diagnosis of post COVID syndrome.
* They have consented to participate in the study
* They have the ability to participate in all aspects of the study.

Exclusion Criteria:

* Pregnant.
* Prior adverse reaction to 14FDG.
* Active implantable medical device e.g. pacemaker, hearing aid implant
* Metallic device e.g. stent, orthopedic hardware in neck
* Using another electronic device at the same time e.g. TENS, mobile phone.
* Any other condition deemed exclusionary by the study principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan T. Hurt, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 12/19/2022 and 03/06/2024, a total of 18 Long Covid patients were found to be eligible to participate in this study through a Long Covid Clinic at a single medical center.
Pre-assignment Details: There was no washout period for this study. After consent, participants were screened, baseline study data were collected and randomized to study groups.
Period: Overall Study
Arm/Group | VNS Treatment | Non-VNS Treatment
Started | 8 | 10
Completed | 8 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VNS Treatment | Non-VNS Treatment | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (10.8) | 46.9 (14.7) | 46.6 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 3 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  NonHispanic/White | 8 | 9 | 17
  Hispanic/White | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Post-COVID Functional Status Score
Description: Measurement is the change in scoring determined through patients' self-reported Post-COVID Functional Status Score survey, which assesses COVID-19 symptom impact on a grading scale of 0 = no limitations to 4 = severe limitations. Thus, higher scores are a worse outcome, and a change indicating an increase is a worsening of functional status.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VNS Treatment | Non-VNS Treatment
Number analyzed (Participants) | 8 | 10
units on a scale | 0.1 (1.0) | 0.3 (0.7)
Statistical Analysis 1: Comparison: VNS Treatment vs Non-VNS Treatment; Test type: Superiority — Groups were compared using Wilcoxon rank sum test; p = 0.544, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in PROMIS Fatigue Scale T Score
Description: Measurement is the change in score determined through patients' self-reported PROMIS Short Form v1.0 - Fatigue 7a. The PROMIS Fatigue Scale assesses 7 items on a scale of 1 (never) to 5 (always). Scale scores were converted to T scores using the published guidelines. A T-score of 50 is the average for the general population with a standard deviation of 10 because calibration testing was performed on a large sample of the general population. A higher PROMIS Fatigue T-score represents more of the concept being measured; thus, an increase in fatigue T score corresponds to more fatigue - which is a worse outcome.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VNS Treatment | Non-VNS Treatment
Number analyzed (Participants) | 8 | 10
units on a scale | -5.4 (11.6) | -1.9 (4.7)
Statistical Analysis 1: Comparison: VNS Treatment vs Non-VNS Treatment; Test type: Superiority; p = 0.292, ANCOVA; ANCOVA was used with the baseline value used as the covariate

ADVERSE EVENTS:
Time Frame: During the 12 weeks of the study treatment period
Arm/Group | VNS Treatment | Non-VNS Treatment
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 2/8 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VNS Treatment (N=8) | Non-VNS Treatment (N=10)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neck Tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT05445427/Prot_SAP_000.pdf